CLINICAL TRIAL: NCT06397716
Title: A Public Health Education and Awareness Initiative on Alcohol Flushing and Alcohol-related Cancer in Asian Communities
Brief Title: Public Health Initiative on Alcohol Flushing
Acronym: AIAC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Stanford Center for Asian Health Research and Education (Unknown)
Responsible Party: Principal Investigator, Kevin Chang, Clinical Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 71764
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Toxicity
Keywords: Alcohol Flushing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotype Revealed (Experimental): Subjects with ALDH2 mutation will be notified of positive genotype results after testing completed.
  Interventions: Genetic: ALDH2 Genotyping
- Gentoype Not-Revealed (Placebo Comparator): Subjects with ALDH2 mutation will not be notified of positive genotype results until after study completed.
  Interventions: Genetic: ALDH2 Genotyping

INTERVENTIONS:
Genetic: ALDH2 Genotyping — Cheek swab for PCR testing of ALDH2 genotype.

SUMMARY:
The overall aim of the study is to raise awareness of alcohol flushing and its health risks to the general population.

The primary objective is to see if spreading awareness of the health risks of alcohol flushing and understanding personalized genotype information will lead to changes in alcohol consumption behavior.

ELIGIBILITY:
Inclusion Criteria:

* Adult age over 18
* Native English speaker

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol Flushing Awareness | Baseline, 1 month, 3 month
  Alcohol flushing reaction awareness questionnaire, scale from 0 to 4, higher score is better outcome
Alcohol Consumption Habits 1 | Baseline, 1 month, 3 month
  Number of days alcohol was consumed in past 30 days
Alcohol Consumption Habits 2 | Baseline, 1 month, 3 month
  Number of days 2 or more drinks of alcohol was consumed in past 30 days
Alcohol Consumption Habits 3 | Baseline, 1 month, 3 month
  Average number of alcohol consumed on days alcohol was consumed
Alcohol Consumption Habits 4 | Baseline, 1 month, 3 month
  Largest number of drinks of alcohol consumed in one sitting

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Chang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No